CLINICAL TRIAL: NCT06856954
Title: The Skin Barrier in Users of Diabetes Devices - Showing the Path to New Way to Prevent and Cure Skin Complications
Brief Title: The Skin Barrier in Users of Diabetes Devices
Acronym: StenoLin
Status: Recruiting | Type: Observational
Sponsor: Jannet Svensson (Other Government)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Jannet Svensson, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: StenoLinskinstudy
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: eczema; lipodystrophy; children; diabetes technology; continous glucose monitor; insulin pump; electric impedance; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Eczema; Lipodystrophy; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes technology (insulin pumps and continuous glucose monitoring) have become standard of care in children with type 1 diabetes. Unfortunately, the attachment of the devices to the skin can provoke injury, irritative or allergic eczema of the skin. Additionally, the continuous insulin infusion often causes sub-cutaneous lipohypertrophy. These occurrences are likely to increase blood glucose fluctuation and impact burden of diabetes. In collaboration with dermatologists, the propose is to investigate the skin microcirculation and skin barrier as well as the subcutaneous tissue when exposed to insulin, occlusion, irritative and allergenic features of the part of device in close contact with the skin. Secondly, investigate the skin barrier and recovery time as a function of time since exposure, type of patches/device and use of preventive strategies like steroids, liquid barrier crème or local anesthetic. To study microcirculation the investgators use Tissue Viability Imaging (TiVI) a non-invasive method using polarization light spectroscopy to count red blood cells thereby saying something about the microcirculation. To investigate skin barrier, the investigators use electric impedance spectroscopy (EIS) which is a non-invasive method sending small electric current of different frequencies through the skin surface. The different frequencies have different properties regarding penetration of cells making it possible to measure the resistance towards each frequency. In this way give a measure of the skin barrier. The last methods investigators are using is ultrasound a non-invasive method that uses sound to show different structures in the subcutaneous tissue, it has been demonstrated to be better than visual inspection to detect lipohypertrophy in the subcutaneous tissue. Lipohypertrophy is often seen in places with repeated infusion/injection of insulin. These investigations are necessary to motivate and guide the development of new materials for diabetes devices and provide clinical guidelines regarding device position and site rotation in order to prevent skin complications from interfering with optimal treatment. This could lead to improved short and long-term outcome in the care of persons with diabetes.

DETAILED DESCRIPTION:
1.2 What is the scientific purpose of the study?

The purpose of the study is to investigate the skin microcirculation and skin barrier as well as the subcutaneous tissue when exposed to insulin, occlusion, irritative and allergenic features of the part of device in close contact with the skin. Secondly, investigate the skin barrier and recovery time as a function of time since exposure, type of patches/device and use of preventive strategies like steroids, liquid barrier crème or local anesthetic

1.3 These are the research questions

1. Do instruction in rotation of insulin pump position using ultrasound improve insulin absorption measured as lower insulin need per kg.
2. Are there detectable differences in measures of skin barrier and micro circulation and visible ultrasound findings comparing the most recent sites of application of devices with regard to material (product) and the attachment time.
3. For how long after diabetes device removal are there visible or measurable changes in the cutaneous and subcutaneous environment of the skin, i.e. how long does the skin need to recover
4. What is the impact on the cutaneous and subcutaneous environment of use of liquid barrier cremes, different patch type, glue removal, different steroid or local anesthetic products
5. Is new device material (e.g. hydrocolloid, silicone or silicone /glycerol) able to impact frequency, extent or recovery time for skin barrier health

Background:

The importance of near normalization of the glucose level in persons with type 1 diabetes (PWD1) is indisputable in securing both short and long-term physical and mental health. Not achieving glycemic targets is associated with an increased risk of short (e.g. hypoglycemic events and hospitalization with diabetic ketoacidosis (DKA)) and long-term complications (e.g. nephropathy, retinopathy, neuropathy and cardiovascular disease). However, achieving strict control is challenging and only a minority reach the current treatment goals even when equipped with insulin pumps and continuous glucose monitoring (CGM/sensor). Modern technology including sensor augmented insulin pumps (SAP) and the new automated insulin delivery systems (AIDs), where CGM values are the basis for an algorithm that adjusts insulin delivery, constitutes an important therapeutic tool that helps PWD1 reach treatment goals and prevents short and long-term complications. The percentage CGM use is correlated with achieving treatment goals. Those using the CGM less than 70% of the time are often excluded from research since in RCT studies the inclusion criteria is using CGM more than 80% of the time and in real-world studies only those with more than 70% CGM data is included. The pre-requisite for using the new technology is a well-functioning infusion set with a subcutaneous tube and CGM attached to the skin.

Eczema and wounds - an obstacle for new technology A major obstacle for using the new technology is the development of eczema and in some cases, an allergy towards the components in the adhesive material or housing of the infusion set (tubing) and CGM. Eczema is seen in 25-33% of children and adults and persists over time, highlighting the lack of proper treatment options. Importantly, skin complications negatively impacts mental health. Shifting to a device with alternative material is seldom an option as the material is often the same across manufactures and although they may contain different acrylates there is a high degree of cross-reaction between acrylates. Nevertheless, for those who develop eczema the beneficial outcomes of insulin pump and CGM treatment outweighs the negative effects, which is why very few stop using the devices leaving little incentive for the manufactures to develop products without allergy provoking substances. The higher costs of alternative material such as silicone or hydrocolloid as well as the possible challenge with adherence adds to the barrier for developing alternatives.

The only known risk factors besides longer-time use (often more than 4 months) is history of atopy making it difficult to predict who would benefit from using preventive strategies like liquid barrier crème or silicone patches underneath to prevent the development of eczema and sensibilization towards e.g. acrylates.

Skin barrier defects may be inherited and mutations in the filaggrin gene contribute to a substantial part, though not all, of those with atopic dermatitis. There is little evidence that persons with type 1 diabetes have higher risk of eczema or atopy than background population since a recent study of the skin barrier showed no difference between PW1D and persons with no diabetes and the investigators could not identify an increased risk of allergic disease in those with type 1 diabetes or vice versa. Therefore, the ingredients/material in the diabetes devices, the closed environment underneath the diabetes devices, mechanical insults or removal practice are the most likely causes of the skin injuries and eczema.

Reuse of the same areas for insulin infusion increases the risk of lipohypertrophy causing impaired absorption of insulin. Ultrasound seems a promising tool for early identification of lipohypertrophy. Reuse also increases skin-stripping when patches are removed repeatedly in the same skin area, increasing the risk of skin barrier defects.

Since an impaired skin barrier increases the risk of contact dermatitis, there is an urgent need for understanding how or whether ingredients/materials in the diabetes devices reaches the skin and may push the skin homeostasis in the wrong direction or damage the epidermal-dermal junction. One study have examined the skin barrier in recent used skin area - showing no recovery within 3 days but clear inflammatory profile at active used skin sites. Further investigations in leasional areas and underneath devices are warranted to shed light on the recovery time and possibility of in differences in skin barrier explain the occurrence of eczema.

Other specific factors have been associated with the development of eczema such as alterations in the natural moisturizing factor (NMF). The investigators found reduced NMF and 2-Pyrrolidone-5-carboxylic acid (PCA) levels in nine adults with long-standing T1D compared to healthy controls, but this applied only for buttock skin. For experimentally induced contact dermatitis and AD, skin barrier impairment has been shown by decreased NMF.

ISPAD guidelines recommend use of proper skin care but also refer to more speculative treatment suggestions such as off-label steroid sprays (e.g., fluticasone) or antiperspirant spray introducing more allergenic substances and a risk of skin atrophy. The available evidence for these recommendations are sparse and only one prospective study has tested the use of proper skin care finding a reduction in wounds/skin injuries but only limited effect on eczema.

The skin barrier can be studied by electric impedance spectroscopy (EIS) a new method that have been shown to detect skin barrier dysfunction in normal looking non-lesional skin of children and predict who is more likely to develop atopic dermatitis. It is able to discriminate between skin without visible changes and healthy skin as well as show a significant increase in EIS that correlated with healing. EIS has also been used to study irritancy from detergents which may be a good surrogate for skin irritation at diabetes treatment sites. Recent studies have been in animal models but historically irritation ( e.g. from sodium laural sulfate has been studied quite extensively with EIS in humans. The microcirculation may be an important marker of skin recovery and skin inflammation seen as hyperemia. Tissue Viability Imaging (TiVI) uses polarization light spectroscopy to study micro vascularization by estimating the red blood cell (RBC) concentration in the skin. The method is very robust and offers instantaneous capturing of data and low variability, though normal values for children and different areas are scarce. The non-invasive properties make EIS and TiVi promising new tools for detecting early signs of skin impairment that could guide how often the individual may reuse site for position of either sensor or infusion set.

The potential healing properties of patches has been studied in some smaller studies where hydrocolloid patches seemed to accelerate healing of the skin and prevent eczema. Material such as silicone or hydrocolloid may be superior to the waterproof and breathable material containing acrylates by reducing the recurrence of eczema and induce optimal condition for fibrinolysis, angiogenesis and wound healing. How use of these type of patches influences the degree of barrier damage, recovery time and normalization as reflected by EIS and TiVi is not investigated although this could potentially support these types of material for future infusion set and sensor patches.

Some children may be reluctant to use new areas for placement of device because of some internal inflexibility and skin complications have been shown to affect quality of life. Therefore, measuring the children's strength and difficulties as well as diabetes specific quality of life may better qualify guidelines of how to help children with skin complications in the future to use new places.

AIM:

The aim of the present study is therefore to investigate the skin micro morphology and skin barrier function using EIS and TiVi in places recently used to attach diabetes devices to investigate differences associated to material and occlusion time as well as recovery time.

And explore the following hypothesis:

Hypothesis:

1. Differences in EIS and TiVi are depending on device type and use of preventive strategies like use of therapeutics (steroid), liquid barrier cremes, glue removal and local anesthetics.
2. EIS and TiVi differ depending on time from removal of the device and material (device type) and use of preventive and treatment strategies
3. Ultrasound detected sub-cutaneous changes depending on reuse of infusion areas (< 4 position in use) and prolonged attachment at the last position (> 3 days *) associates to higher insulin needs per kg and worse glycemic outcome (Higher HbA1c, higher mean glucose and larger glucose variability) *if using extended ware set (EWIS) > 7 days

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 diabetes
* using diabetes device attached to the skin (insulin pump or CGM)

Exclusion Criteria:

* Do not use diabetes device attached to the skin.
* Those unable to read and understand Swedish or English
* impaired cognitive development that may interfere with the ability to answer questionnaires in Swedish/English and/or be reached by phone.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 2 and 17 years of age followed with type 1 diabetes at Crown Princess Victoria Children´s Hospital, Linköping Sweden
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
electric impedance spectroscopy (EIS) | At enrollment and 4 months later at next scheduled ordinary visit
  Electric impedance spectroscopy (EIS) of the skin at last positions of device measured by Nevisense

SECONDARY OUTCOMES:
Tissue Viability Imaging (TiVI) | At enrollment and 4 months later at next scheduled ordinary visit
  Image, that uses polarization light spectroscopy to study micro vascularization by estimating the red blood cell (RBC) concentration in the skin
hyperechogenicity or hypoechogenicity | At enrollment and 4 months later at next scheduled ordinary visit
  Ultrasound detected subcutaneous changes in echogenicity
Time-in-target (TIT: 3.9 - 8 mmol/l) | At enrollment and 4 months later at next scheduled ordinary visit
  Data from continous glucose monitoring (CGM) with TIT the last 30 days before visit
time-below-range (TBR: < 3.9 mmol/l) | At enrollment and 4 months later at next scheduled ordinary visit
  Data from continous glucose monitoring (CGM) with TBR the last 30 days before visit
HbA1c | At enrollment and 4 months later at next scheduled ordinary visit
  HbA1c
Electric impedance spectroscopi (EIS) | At enrollment and 4 months later at next scheduled ordinary visit
  The algorithm derived based on these data from children
eczema | At enrollment and 4 months later at next scheduled ordinary visit
  Visual inspection of the skin and signs of eczema at places where infusions set or CGM devices recently have been placed
wounds | At enrollment and 4 months later at next scheduled ordinary visit
  visual inspection of the last positions for diabetes devices and the occurence of visible wounds
The strength and difficulties questionnaire (SDQ) | At enrollment and 4 months later at next scheduled ordinary visit
  The strength and difficulties questionnaire (SDQ) is a 25 item questionnaire with 5 subscales - a lower score means better strength and less difficulties (range of total score is 0-40). This means a lower score is better.
Diabetes health-related Quality of Life (DISABKIDS) | At enrollment and 4 months later at next scheduled ordinary visit
  Diabetes health-related Quality of Life (Disabkids) questionnaire with 10 items and 2 subscales - total score range is from 0 to 40 and higher score means a more negative impact from diabetes on quality of life and therefore worse

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Svensson, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Crown Princess Victoria Children´s Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Depending on Swedish law, if possible without hampoering GDPR the data will be shared